CLINICAL TRIAL: NCT04976985
Title: The Efficacy of Osteopathic Manipulative Treatment on Decreasing the Severity of Migraine Headaches
Brief Title: Osteopathic Manipulative Treatment and Migraine Headaches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-106
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Chronic Migraine; Migraine Disorders; Headache Disorders; Headache, Migraine
Keywords: OMT; Osteopathic Manipulative Therapy; Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache Disorders; Headache | interventions — Manipulation, Osteopathic; Standard of Care

STUDY DESIGN:
Intervention Model Description: Interventional group: 70 patients with chronic migraine who consent to OMT will receive four standardized osteopathic manipulative treatments over the course of twelve weeks. MIDAS and HIT-6 Questionnaires will be obtained at time of consent prior to first treatment and again at the conclusion of treatment period of twelve weeks.
  Control Group: 70 patients with the diagnosis of migraine headache will complete a MIDAS and HIT-6 questionnaire at week 0 and week 12 on standard of care for migraine treatment. A new prophylactic medication may be started at time of initial questionnaires and the patient can be on up to two prophylactic medications, with no changes during the 12 week period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group receiving Osteopathic Manipulative Therapy (OMT) (Experimental): 70 patients with chronic migraine who consent to OMT will receive four standardized osteopathic manipulative treatment protocol over the course of twelve weeks at week 0,2,6,10. MIDAS and HIT-6 Questionnaires will be obtained at time of consent prior to first treatment and again at the conclusion of treatment period of twelve weeks.
  Interventions: Procedure: Osteopathic Manipulative Therapy (OMT)
- Control Group with Standard of Care (Other): 70 patients with the diagnosis of migraine headache who are receiving the standard of care medications will complete a MIDAS and HIT-6 questionnaire at week 0 and week 12. A new prophylactic medication may be started at time of initial questionnaires and the patient can be on up to two prophylactic medications, with no changes during the 12 week period.
  Interventions: Other: Standard of care

INTERVENTIONS:
Procedure: Osteopathic Manipulative Therapy (OMT) — Osteopathic Manipulative Therapy (OMT) is a non-pharmacological, noninvasive form of manual medicine. Osteopathic physicians receive special training in the musculoskeletal system to detect somatic dysfunction. Osteopathic physicians then move a patient's muscles and joints using techniques that include stretching, gentle pressure and resistance to improve muscle tonicity, treat structural abnormalities, relieve joint restriction, and decrease activation of the pain proprioception pathway.
  OMT Standardized Protocol A:
  1. Occipital- Alanto release
  2. Muscle energy and soft tissue to mid trapezius muscle
  3. Muscle energy to cervical spine in all three planes of flexion/extension, rotation and side bending
  4. Screening for tender points of C2-C6 at transverse and spinous processes and treatment with counterstain if tender point identified
  5. Soft tissue to cervical paraspinal muscles
  6. Myo-fascial release of frontal forehead
  7. CV4 cranial technique
  Other Names: OMT
  Arms: Interventional Group receiving Osteopathic Manipulative Therapy (OMT)
Other: Standard of care — Receiving standard of care for migraine headaches with pharmacological medications, with no more than two prophylactic medications during the study period. Participants may also take abortive migraine medications.
  Arms: Control Group with Standard of Care

SUMMARY:
In this study the investigators hypothesize, that Osteopathic Manipulative Therapy (OMT) will reduce migraine disability and severity scores when compared to standard of care including prophylactic pharmacological agents with treatment over 12 week time frame. The investigators aim to decrease severity and disability of migraine by utilizing Osteopathic Manipulative Therapy. This would ultimately reduce the utilization of office or emergency department visits, decrease the large economic burden the United States faces for migraine patients as well as improve quality of life for the 3 million chronic migraine patients.

DETAILED DESCRIPTION:
According to the American Headache Society, Migraine headaches affect one billion people worldwide. In the United States, one in five women and one in sixteen men suffer from migraine headaches. Migraine is the sixth most disabling illness in the world. More than four million people have chronic daily migraines with at least 15 migraines per month. More than 90% of sufferers are unable to work or function normally during their migraine attacks. Unlike many other chronic diseases, migraine affects otherwise healthy, young and middle aged people. Headache accounts for the fourth or fifth most common reason for emergency department visits and the economic burden of migraine reaches $78 billion dollars per year.

Osteopathic Manipulative Therapy (OMT) is a non-pharmacological, non-invasive form of manual medicine. Headache has been shown to be associated with impairment of autonomic nervous system including autonomic nuclei responsible for pain perception. It has also been shown through research that persons with a migraine episode are known to release high levels of the pro-inflammatory agents, prostaglandins, dopamine and serotonin. The effect of OMT on headache can be two fold: First, by increasing parasympathetic tone, and second, by inhibiting pro-inflammatory substances. Therefore, OMT could theoretically counter balance both the release of pro-inflammatory markers as well as the autonomic nervous system leading to improved clinical outcomes. These outcomes include: decreasing patients' severity and frequency of their migraine headache, which, ultimately could improve subjects' productivity to society and decrease the economic burden of migraine sufferers.

Historically, OMT was believed to worsen migraine headaches, this study is being conducted to learn about how Osteopathic Manipulative Therapy can help migraine patients. Subjects receiving OMT could benefit from improved quality of life by reducing subject's severity and frequency of their migraine headache, which could improve their productivity to society and decrease the economic burden of migraine headaches. This could provide information to make Osteopathic Manipulative Therapy an acknowledged alternative therapy to improve quality of life for 3 million chronic migraine sufferers.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-50
2. Gender: Male and Female
3. ICD 10 code of migraine with or without aura (G43.0, G43.1, G43.70, G43.71)
4. No change in prophylactic medication for both control and intervention group
5. No physical therapy for headaches, neck pain or for trapezius muscle during 12 weeks for both control and intervention group

Exclusion Criteria:

1. Previous Surgery to neck or cranium, history of previous stroke
2. More than two daily prophylactic pharmacologic agents used for the indication of Migraine headache
3. Active cancer
4. Receiving BOTOX® for migraines or treatment within the last 4 months
5. If patient has contraindications for OMT for the intervention group such as clinical signs of fractures in cervical spine, ligament instability, or severe vertebral artery stenosis
6. If patient is poor candidate for OMT in intervention group such as the patient is unable to follow commands.
7. Seizure disorder or recent head trauma
8. Pregnant or become pregnant during the treatment period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in the Migraine Disability Test (MIDAS) score in the OMT interventional group compared to control group. | 12 weeks
  Reduction in the Migraine Disability Test (MIDAS) score and level of disability per the MIDAS score scoring system:
  MIDAS Grade I (Little to no disability): 0-5 MIDAS Grade II(Mild Disability): 6-10 MIDAS Grade III (Moderate Disability): 11-20 MIDAS Grade IV (Severe Disability): 21+
  minimum score: 0 maximum score: 21+ (no maximum)
Reduction in the Headache Impact Test (HIT-6) score in OMT intervention group compared to control group. | 12 weeks
  Reduction in the Headache Impact Test (HIT-6) score per the scoring system:
  Little or no impact: 49 or Less Some impact: 50-55 Substantial Impact: 56-59 Severe Impact: 60-78
  minimum score: 36 Maximum score: 78

SECONDARY OUTCOMES:
Headache Days | 12 weeks
  Reduction in the number of headache days over 12 weeks
Pain scale | 12 weeks
  Reduction in the pain scale (1-10) for migraine headaches

CONTACTS AND LOCATIONS:
Overall Officials: Abby Rhoads, DO, Principal Investigator — St. Luke's Hospital and Health Network, Pennsylvania
Locations (1):
- St. Luke's University Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burch R, Rizzoli P, Loder E. The Prevalence and Impact of Migraine and Severe Headache in the United States: Figures and Trends From Government Health Studies. Headache. 2018 Apr;58(4):496-505. doi: 10.1111/head.13281. Epub 2018 Mar 12. PMID 29527677
- [Background] Carnes D, Mars TS, Mullinger B, Froud R, Underwood M. Adverse events and manual therapy: a systematic review. Man Ther. 2010 Aug;15(4):355-63. doi: 10.1016/j.math.2009.12.006. Epub 2010 Jan 22. PMID 20097115
- [Background] Cerritelli F, Lacorte E, Ruffini N, Vanacore N. Osteopathy for primary headache patients: a systematic review. J Pain Res. 2017 Mar 14;10:601-611. doi: 10.2147/JPR.S130501. eCollection 2017. PMID 28352200
- [Background] Voigt K, Liebnitzky J, Burmeister U, Sihvonen-Riemenschneider H, Beck M, Voigt R, Bergmann A. Efficacy of osteopathic manipulative treatment of female patients with migraine: results of a randomized controlled trial. J Altern Complement Med. 2011 Mar;17(3):225-30. doi: 10.1089/acm.2009.0673. Epub 2011 Mar 8. PMID 21385086
- [Background] McReynolds TM, Sheridan BJ. Intramuscular ketorolac versus osteopathic manipulative treatment in the management of acute neck pain in the emergency department: a randomized clinical trial. J Am Osteopath Assoc. 2005 Feb;105(2):57-68. PMID 15784928
- [Background] Zein-Hammoud M, Standley PR. Modeled Osteopathic Manipulative Treatments: A Review of Their in Vitro Effects on Fibroblast Tissue Preparations. J Am Osteopath Assoc. 2015 Aug;115(8):490-502. doi: 10.7556/jaoa.2015.103. PMID 26214822
- [Background] Francesco Cerritelli, et al. Is osteopathic manipulative treatment effective in migraine?. International Journal of Osteopathic Medicine. March 2013Volume 16, Issue 1, Pages e1-e2.
- See also: AOA - What is Osteopathic Medicine — https://osteopathic.org/what-is-osteopathic-medicine/osteopathic-manipulative-treatment/